CLINICAL TRIAL: NCT04926766
Title: Super Hypofractionated Irradiation for Whole Breast Treatment: a Prospective, Single-arm Trial
Brief Title: Super Hypofractionated Irradiation for Whole Breast Treatment
Acronym: SHIFT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, JIAYI CHEN, Chief of Department of Radiation Oncology, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHF-WBI
Record Dates: First submitted 2021-06-09; First posted 2021-06-15 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer
Keywords: Whole breast irradiation; IMRT; Super Hypofractionated radiotherapy; Super Hypofractionated irradiation to tumor bed boost
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SHF-WBI (Experimental): Patients with an indication for whole breast irradiation will receive 5.2 Gy in 5 fractions to whole breast and a sequential tumor bed boost of 5.2 Gy in 2 fractions at the discretion of radiation oncologist
  Interventions: Radiation: External Beam radiotherapy using IMRT technique

INTERVENTIONS:
Radiation: External Beam radiotherapy using IMRT technique — 2600cGy/ 5 fractions / 1 weeks to ipsilateral whole breast and a sequential tumor bed boost of 5.2 Gy in 2 fractions at the discretion of radiation oncologist

SUMMARY:
The purpose of this trial is to investigate the safety and efficacy of super hypofractionated whole breast irradiation (SHF-WBI) in breast cancer patients treated with breast conserving surgery. Eligible breast cancer patients will be followed for at least 5 years to evaluate the acute and late radiation-induced toxicities, locoregional recurrence, distant metastasis, death, contralateral breast cancer and quality of life.

DETAILED DESCRIPTION:
Eligible breast cancer patients will receive SHF-WBI of 5.2 Gy in 5 fractions to ipsilateral whole breast within one week and a sequential tumor bed boost of 5.2 Gy in 2 fractions at the discretion of the radiation oncologist. All patients are treated with intensity modulated radiation therapy (IMRT) technique. The primary endpoint is ≥2 grade any acute radiation induced toxicity event. Patients will be followed for at least 5 years to evaluate the acute and late radiation-induced toxicity, locoregional recurrence, distant metastasis, death and quality of life.

Calculation of the required number of cases based on an alpha of 0.05 and a power of 80% with a maximal tolerable toxicity difference of 10% during and within 6 months after SHF-WBI comparing to hypofractionated whole breast irradiation(40-42.5Gy/15-16Fx) and lost rate of follow up of 10%. In total 217 patients are needed to be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Aged ≥18 years old
* breast conservation surgery
* unilateral histologically confirmed invasive breast carcinoma or Ductal Carcinoma In Situ (DCIS)
* For patients with invasive breast cancer，negative axillary lymph nodes or micrometastasis only
* Karnofsky Performance Status ≥80, and Life expectancy of >5 years
* Histologically negative surgical margin for invasive breast carcinoma or a minimum negative margin width of ≥ 3mm for DCIS
* Surgery wound healed without infection
* ER (estrogen-receptor), PR (progesterone-receptor), HER2 (human epidermal growth factor receptor 2) and Ki67 testing can be performed on the primary breast tumor
* Female patients of child-producing potential must agree to use effective contraception for up to 1 month before study treatment and the duration of study participation

Exclusion Criteria:

* Histological involvement of supraclavicular lymph node
* Histologically or radiologically confirmed involvement of ipsilateral internal mammary lymph nodes
* Pregnant or lactating women
* Severe non-neoplastic medical comorbidities
* Diagnosis of non-breast malignancy within 5 years preceding enrollment (excluding lobular carcinoma in situ, basal cell carcinoma of the skin, carcinoma in situ of skin and carcinoma in situ of the cervix, Pulmonary adenocarcinoma in situ，which are permitted).
* simultaneous contralateral breast cancer
* Previous radiotherapy to the neck, chest and/or ipsilateral axillary region
* Active collagen vascular disease
* Definitive histological or radiologic evidence of distant metastatic disease
* Evidence of T4 disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Estimated)
Dates: Start 2021-01-23 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2028-07-10 (Estimated)

PRIMARY OUTCOMES:
Cumulative complication rate of ≥Grade 2 Acute Radiation-induced Toxicity | 6 months
  Within time from the beginning of radiotherapy to 6 months after completion of radiotherapy, any acute radiation induced toxicities will be assessed and recorded using Common Terminology Criteria for Adverse Events (CTCAE) 5.0.

SECONDARY OUTCOMES:
Cumulative complication rate of ≥Grade 2 Late Radiation-induced Toxicity | 5 years
  Within time from 6 months after completion of radiotherapy to 5 years after completion of radiotherapy, any late toxicity will be assessed and recorded using the Radiation Therapy Oncology Group (RTOG) /European Organization for Research on Treatment of Cancer (EORTC) Late Radiation Morbidity Scoring Schema and CTCAE 5.0
Number of Participants with excellent or good Cosmetic outcomes following breast conserving surgery-Harvard/ NSABP/RTOG scoring scale | 6 months
  The cosmetic outcomes will be evaluated at 6 months after last fractions. The cosmetic outcomes are evaluated based on the Allegheny General Modification of the Harvard/National Surgical Adjuvant Breast and Bowel Project (NSABP)/RTOG scoring scale which graded patients into the following four classifications: excellent, when compared to the untreated breast, there is a minimal or no difference in the size or shape of the treated breast; good, slight difference in the size or shape of the treated breast; fair, obvious difference in the size or shape of the treated breast; and poor, marked change in the size or shape of the treated breast
Number of Participants with excellent or good Cosmetic outcomes following breast conserving surgery-Harvard/ NSABP/RTOG scoring scale | 5 years
  The cosmetic outcomes will be evaluated at 5 years after last fractions. The cosmetic outcomes are evaluated based on the Allegheny General Modification of the Harvard/National Surgical Adjuvant Breast and Bowel Project (NSABP)/ RTOG scoring scale which graded patients into the following four classifications: excellent, when compared to the untreated breast, there is a minimal or no difference in the size or shape of the treated breast; good, slight difference in the size or shape of the treated breast; fair, obvious difference in the size or shape of the treated breast; and poor, marked change in the size or shape of the treated breast
Locoregional recurrence | 5 years
  any first recurrence confirmed by histology or cytology within the ipsilateral chest wall and/or regional nodes area(including supraclavicular, infraclavicular or internal mammary lymph nodes)
Distant metastasis free survival (DMFS) | 5 years
  The time from the date of enrollment to any recurrence of tumor at distant sites or death from any cause
Invasive recurrence-free survival (IRFS) | 5 years
  The time from the date of enrollment to any invasive recurrence of tumor or death from any cause
Overall survival | 5 years
  The time from the date of enrollment to the date of death from any cause

OTHER OUTCOMES:
Quality of Life-EORTC QLQ-C30 | 6 months
  Quality of life will be assessed before radiotherapy and 6 months after last fractions using self administered questionnaire EORTC QLQ-C30
Quality of Life-EORTC QLQ-C30 | 5 years
  Quality of life will be assessed before radiotherapy and 6 months after last fractions using self administered questionnaire EORTC QLQ-C30
Quality of Life-EORTC QLQ-BR23 | 6 months
  Quality of life will be assessed before radiotherapy and 6 months after last fractions using self administered questionnaire EORTC QLQ-BR23
Quality of Life-EORTC QLQ-BR23 | 5 years
  Quality of life will be assessed before radiotherapy and 6 months after last fractions using self administered questionnaire EORTC QLQ-BR23

CONTACTS AND LOCATIONS:
Overall Officials: Jiayi Chen, PhD, MD, Study Chair — Ruijin Hospital Affiliated to Shanghai Jiaotong University School of Medcine; Lu Cao, PhD, MD, Principal Investigator — Ruijin Hospital Affiliated to Shanghai Jiaotong University School of Medcine
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No